CLINICAL TRIAL: NCT05209139
Title: Acute Effects of Beetroot Juice Ingestion on Neuromuscular Performance and Match-play Demands in Elite Female Hockey Players.
Brief Title: Beetroot Juice Ingestion Effects on Field Hockey Performance.
Acronym: BEETHOCKEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: University of Alcala (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidad Francisco_Vitoria
Record Dates: First submitted 2022-01-14; First posted 2022-01-26 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Nitrates; Hockey
Keywords: dietary supplements; sports nutrition; field hockey; female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot supplementation (Experimental): Acute beetroot juice supplementation
  Interventions: Dietary Supplement: Beetroot juice; Dietary Supplement: Beetroot juice placebo
- Placebo supplementation (Placebo Comparator): Acute placebo supplementation
  Interventions: Dietary Supplement: Beetroot juice; Dietary Supplement: Beetroot juice placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice — One serving 70 mL of beetroot juice (6.4 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.
Dietary Supplement: Beetroot juice placebo — One serving 70 mL of beetroot juice placebo (0.04 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.

SUMMARY:
Scientific evidence supports that only a few dietary supplements have reported good evidence for improving sports performance, between we can mention beetroot juice supplementation with doses > 5 mmol of NO3-. In this randomized placebo-controlled study, we investigated the effects of BJ acute supplementation in improving neuromuscular performance and match-play demands in female field hockey players.

DETAILED DESCRIPTION:
Beetroot juice supplementation has demonstrated good evidence for improving sports performance, however, benefits in team sports, especially in female athletes, are underrepresented. In this randomized placebo-controlled study, we investigated the effects of beetroot juice acute supplementation in improving neuromuscular performance and match-play demands.Testing sessions will comprise a neuromuscular test battery consisting of a countermovement jump (CMJ), isometric handgrip strength, 20-m sprint and repeated sprint ability test, followed by a 20-minute simulated field hockey Physical match activity (distances, speeds, accelerations and decelerations) will be monitored in real-time using an inertial tracking system

ELIGIBILITY:
Inclusion Criteria:

* Elite female field hockey players (playing in First Field Hockey Division).
* More than 8 years of field hockey training experience.

Exclusion Criteria:

* Concurrently participating in other studies.
* Contraindications associated to beetroot ingestion.
* Health problems or musculoskeletal injuries 6 months previous to study realization

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in simulated field hockey match demands (m/min) | 1 week
  Using a global position system (GPS)
Changes in repeated-sprint-ability test (s) | 1 week
  Time to complete the modified repeated sprint ability test using photocell timing gates

SECONDARY OUTCOMES:
Changes in sprint time (s) | 1 week
  Time to complete 20-m sprints using photocell timing gates
Changes in maximal jump height (cm) | 1 week
  Maximal jump height using a contact platform
Changes in maximal isometric handgrip strength (N) | 1 week
  Using a hand-held dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez-Samanes A, Perez-Lopez A, Morencos E, Munoz A, Kuhn A, Sanchez-Migallon V, Moreno-Perez V, Gonzalez-Frutos P, Bach-Faig A, Roberts J, Dominguez R. Beetroot juice ingestion does not improve neuromuscular performance and match-play demands in elite female hockey players: a randomized, double-blind, placebo-controlled study. Eur J Nutr. 2023 Apr;62(3):1123-1130. doi: 10.1007/s00394-022-03052-1. Epub 2022 Nov 19. PMID 36401662